CLINICAL TRIAL: NCT05629819
Title: Effect of Early Non-invasive Phrenic Nerve Stimulation on Weaning in Mechanically Ventilated Patients：A Multicenter, Randomized Controlled Study
Brief Title: Effect of Early Non-invasive Phrenic Nerve Stimulation on Weaning in Mechanically Ventilated Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Bing Sun (Other)
Responsible Party: Sponsor-Investigator, Bing Sun, professor of treatment, Beijing Chao Yang Hospital
Organization: Beijing Chao Yang Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: PNS in MV patients
Record Dates: First submitted 2022-11-11; First posted 2022-11-29 (Actual); Last update posted 2024-03-26 (Actual); Status verified 2024-03

CONDITIONS: Mechanical Ventilation; Weaning
Keywords: phrenic nerve stimulation; diaphragm function

STUDY DESIGN:
Who Masked: Participant
Masking Description: Patients enrolled in the study were unaware of the study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PNS group (Experimental): In addition to conventional respiratory therapy and pulmonary rehabilitation, neuromuscular electrical stimulator was used for PNS
  * Device Settings Strength: Maximum current tolerated by the patient (0-100mA, commonly used below 13mA) ； Stimulation time: 1.0s; Frequency: 40Hz;
  * Location: The stimulation electrodes were attached to the left and right sides of the neck under the outer margin of the sternocleidomastoid muscle 1/3; The reference electrodes were attached to the surface of both pectoralis major muscles.
  * Treatment frequency: 30 at a time, Bid, until withdrawal/death/for 4 weeks.
  Interventions: Device: Non-invasive phrenic nerve stimulation
- conventional group (No Intervention): * conventional respiratory therapy and pulmonary rehabilitation, including airway management, early activity, and respiratory muscle training.
  * No intervention

INTERVENTIONS:
Device: Non-invasive phrenic nerve stimulation — Some studies have shown that PNS can relieve diaphragmatic atrophy and reverse diaphragmatic dysfunction.
  Arms: PNS group

SUMMARY:
the early application of non-invasive PNS in MV patients can increase the number of days without mechanical ventilation, delay disuse phrenic atrophy, and improve the strength of inspiratory muscle.

DETAILED DESCRIPTION:
A prospective randomized controlled study included 104 patients with MV who met inclusion criteria in multiple hospital ICU units and were randomly divided 1:1 into PNS and conventional groups. The PNS group received neuromuscular electrical stimulation in addition to routine airway management, early activity and respiratory muscle training. It was verified that early non-invasive PNS could increase the number of days without mechanical ventilation for 28 days, delay disused diaphragm atrophy and improve inspiratory muscle strength.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18years and ≤80years;
* MV time ≤48h;
* MV duration is expected to be ≥72h;
* The sternocleidomastoid region and pectoralis major region were completely exposed.
* Patients or family members are willing to sign informed consent and participate in the study.

Exclusion Criteria:

* There are contraindications to PNS in vitro (Pneumothorax, active tuberculosis, pleural adhesions, installation of pacemakers and defibrillators, etc.);
* Neuromuscular disease (myasthenia gravis, etc.) or known anatomical abnormalities of the diaphragm;
* ECMO status;
* Hemodynamic instability;
* Uncorrected arrhythmias;
* Be pregnant;
* Clinical end-stage and palliative care patients.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Ventilator-free days | 28 days

SECONDARY OUTCOMES:
mechanical ventilation days | 28 days
re-intubation rate | 28 days
ICU mortality | 28 days
60/90-day survival rate | 28 days
Maximal Inspiratory Pressure | up to 28 days
Diaphragm thickness | up to 28 days
diaphragm thickening fraction | up to 28 days
Transdiaphragmatic Pressure | up to 28 days

OTHER OUTCOMES:
The incidence of adverse events | up to 28 days
Medical expenses | through study completion, an average of 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Bing Sun, MD, Principal Investigator — Beijing Chao Yang Hospital
Locations (1):
- Bing Sun, Beijing, Beijing Municipality, China